CLINICAL TRIAL: NCT02663765
Title: Impact of Lack of Antenatal Care in Primiparas on Maternal and Perinatal Outcomes
Brief Title: Lack of Antenatal Care in Primiparas
Acronym: ANC
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Lecturer, Assiut University
Other Study IDs: ANC
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Antenatal Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Antenatal care is a key strategy for reducing maternal and neonatal morbidity and mortality rate because adequate utilization of antenatal health care services is associated with improved maternal and neonatal health outcomes. The trend of maternal mortality in developing countries has been increasing and various international organizations have reported that an important factor related to maternal and infant mortality has been linked to lack of antenatal care. According to Federal Ministry of Health, some of the dangers of pregnancy and childbirth can be avoided if the pregnant woman attends antenatal regularly. In order to decrease these mortality rates, regular antenatal care has to be instituted or reinforced which can only be achieved through identifying factors causing poor utilization of antenatal care services

ELIGIBILITY:
Inclusion Criteria:

* Women who agree to participate in the study
* Primipara.

Exclusion Criteria:

* Multipara.
* Women who refuse to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: primiparas who will be delivered in Assiut Women Health Hospital
Sampling Method: Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
number of morbidity cases due to lack of antenatal care | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No